CLINICAL TRIAL: NCT06395532
Title: Integrated Pulmonary Index as a Predictor of Respiratory Compromise in Critically Ill Patients: A Prospective, Observational Study
Brief Title: Integrated Pulmonary Index as a Predictor of Respiratory Compromise in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Professor, Ain Shams University
Other Study IDs: FMASU MS 136/2024.
Record Dates: First submitted 2024-04-23; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Respiratory compromise (RC) group
  Interventions: Other: Observetional
- Non respiratory compromise (RC) group
  Interventions: Other: Observetional

INTERVENTIONS:
Other: Observetional — After admission to the ICU, patients will be continuously monitored with ICU standard monitoring in addition to IPI using (Capnostream™ Medtronic). IPI will be recorded after transfer to the ICU, as well as at 2, 6, 12, 18 and 24 hours.

SUMMARY:
The integrated pulmonary index (IPI) is a newly developed index for respiratory monitoring. However, there is limited evidence on its effectiveness and usefulness in critically ill patients. The purpose of this study is to evaluate the clinical relevance of the IPI as a predictor of respiratory compromise in critically ill patients.

DETAILED DESCRIPTION:
Recent developments aim to use multiple parameters to detect AREs. Application of smart algorithms that combine individual physiological variables into one index may increase the ability to detect a true adverse respiratory event while avoiding false alarms and limiting alarm fatigue.

An example of such a multiparameter index is the Integrated Pulmonary Index or IPI™, which integrates oxygen saturation (SpO2), respiratory rate (RR), end-tidal PCO2 (PETCO2) and heart rate (HR) into a single integer value of 1-10 that represents adequacy of respiratory condition of the patient using a fuzzy logic inference mathematical model; scores ≥ 8 points are within normal range and those ≤ 4 points suggest requirement of interventions.

The IPI algorithm summarizes the state of ventilation and oxygenation at the point in time. Previous studies reported that IPI correlated with respiratory physiological parameters of patients undergoing sedation for surgeries or for colonoscopy.

Up to our knowledge, the clinical relevance of the IPI as a predictor of respiratory compromise in critically ill patients has not been discussed before.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients aged 18 years or older of both genders admitted to the intensive care unit

Exclusion Criteria:

* Age < 18 years' old
* Morbid obesity
* Mechanical ventilation
* Hemodynamic instability.
* Thoracotomy and cardiac surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients will receive the standard care, according to the usual standard clinical practice at the institution. After admission to the ICU, patients will be continuously monitored with ICU standard monitoring in addition to IPI using (Capnostream™ Medtronic). IPI will be recorded after transfer to the ICU, as well as at 2, 6, 12, 18 and 24 hours. Any respiratory, hemodynamic events or interventions will be recorded by the ICU nurses who will be blinded for the study.Demographic ( age, gender, BMI, co morbidities), clinical, laboratory, and outcomes data will be obtained from the medical records. Routine laboratory tests were done for all patients, including CBC, C-reactive protein, renal profile, coagulation profile and liver profile.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-11-16 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Respiratory Failure | 6 months
  1. Hypoxia
  2. Hypercapnia

SECONDARY OUTCOMES:
Complications | 6 months
  1. The onset of Mechanical ventilation
  2. The Duration of Mechanical ventilation
  3. lCU length of stay
  4. Hospital length of stay 5-28 days mortality